CLINICAL TRIAL: NCT01579721
Title: Prospective Randomized Study of Single Incision Laparoscopic Surgery Versus Conventional Laparoscopic Surgery for Rectal Cancer
Brief Title: Prospective Randomized Study of SILS Versus CLS for Rectal Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Katrine Kanstrup Aslak, MD, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SILS rectal cancer
Record Dates: First submitted 2012-04-16; First posted 2012-04-18 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Rectal Cancer; Adenocarcinoma
MeSH Terms: conditions — Rectal Neoplasms; Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SILS-group (Experimental): 20 patients undergoing Single Incision Laparoscopic Surgery
  Interventions: Procedure: Single Incision Laparoscopic Surgery
- CLS-group (No Intervention): 20 patients undergoing Conventional Laparoscopic Surgery for rectal cancer

INTERVENTIONS:
Procedure: Single Incision Laparoscopic Surgery — Single incision laparoscopic surgery for rectal cancer
  Arms: SILS-group

SUMMARY:
Background: Single-port laparoscopic surgery is emerging as a method to improve morbidity and cosmetic benefits of conventional laparoscopic surgery and minimize the surgical trauma. However, the feasibility of this procedure in rectal surgery has not been determined yet. The aim of this study is to evaluate our initial experience using single port access in laparoscopic rectal surgery.

Design: randomized, prospective clinical study Patients: 40 patients

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age.
* ASA I-III.
* Tumor-location: maximum 15 cm from the anal verge.
* No involvement of neighbouring organs.
* No distant metastasis.

Exclusion Criteria:

* Linguistic, physical or psychological barriers precluding oral and written consent.
* History of intestinal surgery (excl. appendectomy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
morbidity | 30 days
  The purpose of this study is to compare 30-days postoperative morbidity between the two groups

SECONDARY OUTCOMES:
immunology | 72 hours postoperatively
  to compare results of blood-samples (C-reactive protein, leucocyte-count and interleukin-6) 72 hours postoperatively between the two groups
postoperative outcome | 5 days postoperatively
  to compare postoperative results (postoperative pain, time to bowel function, time to regain full diet and mobilisation) between the two groups.
oncology | 30 days
  Comparison of the oncological results (quality of specimen, completeness of mesorectal fascia, circumferential resection margin, number of harvested lymphnodes, TNM-classification) between the two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroentestinal Surgery, Hvidovre Hospital, Hvidovre, Denmark

REFERENCES:
- [Derived] Bulut O, Aslak KK, Levic K, Nielsen CB, Romer E, Sorensen S, Christensen IJ, Nielsen HJ. A randomized pilot study on single-port versus conventional laparoscopic rectal surgery: effects on postoperative pain and the stress response to surgery. Tech Coloproctol. 2015 Jan;19(1):11-22. doi: 10.1007/s10151-014-1237-6. Epub 2014 Nov 8. PMID 25380743